CLINICAL TRIAL: NCT03067038
Title: Single Incision Versus Three Port Laparoscopic Cholecystectomy in Symptomatic Gallstones: A Prospective Randomized Study
Brief Title: Single Incision Versus Three Port Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, Lecturer of GIT surgery and laparoendoscopy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU
Record Dates: First submitted 2016-11-25; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single incision LC (Active Comparator): Single incision laparoscopic cholecystectomy (SILC) performed through a single infra-umbilical incision using a single port device or three ports closely placed.
  Interventions: Device: Single incision laparoscopic cholecystectomy
- Three port LC (Sham Comparator): Three port laparoscopic cholecystectomy (TPLC) performed through three different placed trocars
  Interventions: Device: Three port laparoscopic cholecystectomy

INTERVENTIONS:
Device: Single incision laparoscopic cholecystectomy — Laparoscopic cholecystectomy with single port device
  Arms: Single incision LC
Device: Three port laparoscopic cholecystectomy — Laparoscopic cholecystectomy with three port
  Arms: Three port LC

SUMMARY:
Laparoscopic cholecystectomy (LC) became the standard treatment for symptomatic gallbladder disease. Single incision laparoscopic surgery (SILS) was developed with the aim of reducing the invasiveness of conventional laparoscopy. The aim of this study was to compare the clinical outcome of single-incision laparoscopic cholecystectomy (SILC) with three port laparoscopic cholecystectomy (TPLC).

DETAILED DESCRIPTION:
From February 2014 to September 2016, patients with symptomatic cholecystolithiasis at two university hospitals (Sohag University and Qena University hospitals) were enrolled in this study.

The number of patients needed was calculated. Considering a power of 80% and reliability of 0.05, the investigator found that 76 patients should be present in each group. The study was started with 275 patients for the possible loss of patients and data during the study. Eligible patients (206 patients) were randomly divided equally into two groups (Group 1; SILC, Group 2; TPLC) according to a computer-generated random numbers. Of 103 patients allocated to intervention in each group, 14 patients were excluded from SILC group and 5 patients from TPLC group, and the remaining 89 & 98 patients in SILC & TPLC group respectively were included in the study.

Routine investigations and surgical fitness were done in all cases. Patient demographics, BMI, ASA score, indication for cholecystectomy, operative time, estimated blood loss, success and conversion rate, postoperative pain score, postoperative analgesia requirement, morbidity and mortality, length of hospital stay, and patient cosmetic satisfaction were recorded.

A fixed analgesia protocol with intravenous non-narcotic (ketorolac tromethamine 30 mg) was used twice daily. An opioid (pethidine Hcl 50 mg) was added when the pain cannot be tolerable. Postoperative pain was evaluated according to a visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain) on the postoperative sixth hour (VAS-6H) and on postoperative day one (VAS-24H). Patient cosmetic satisfaction was recorded at one month follow-up visit on a scale from 1 (worst) to 10 (best). Patients were shown the same photograph of a right sub-costal (Kocher) incision which was rated 0 on the cosmetic scale and were asked to rate their satisfaction based on the previous observation. The study protocol was approved by the local ethical committee. Also, a written informed consent was obtained from all patients' prior recruitment to study.

ELIGIBILITY:
Inclusion Criteria:

1. preoperative diagnosis of symptomatic gallstones
2. age from 20 to 60 years,
3. American Society of Anesthesiologists (ASA) grade I, II or III,
4. agreement to complete the study requirement.

Exclusion Criteria:

1. patients with contraindication to laparoscopy,
2. suspected Mirizzi syndrome,
3. choledocholithiasis,
4. hepatobiliary malignancy,
5. previous upper abdominal surgery,
6. previous mesh repair of an umbilical hernia,
7. long-term anticoagulant treatment,
8. pregnant female
9. stone more than 2 cm in preoperative ultrasonography.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
postoperative pain, visual analogue scale (VAS) | at 6 hours
  Postoperative pain was evaluated according to a visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain) on the postoperative hour six (VAS-6H).
postoperative pain, visual analogue scale (VAS) | at 24 hours
  Postoperative pain was evaluated according to a visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain) on the postoperative day one (VAS-24H).

SECONDARY OUTCOMES:
operative duration | From introduction of first trocar to the recovery of patient, up to 10 hours
post operative opioid requirements (questioner) | 24 hours
lenght of hospital stay | from recovery of anaesthesia to discharge of patient, up to 4 days
cosmetic satisfactions (aesthetic scale) | one month
  Patient aesthetic satisfaction was recorded at one month follow-up visit on a scale from 1 (worst) to 10 (best). Patients were shown the same photograph of a right sub-costal (Kocher) incision which was rated 0 on the aesthetic scale and were asked to rate their satisfaction based on the previous observation.

IPD SHARING:
Plan to Share IPD: No